CLINICAL TRIAL: NCT03380390
Title: Multicenter, Open-Label, Interventional Study on the Safety and Tolerability of Oxymetazoline and Energy-Based Therapy in Subjects With Rosacea
Brief Title: Safety and Tolerability of Oxymetazoline and Energy-Based Therapy in Participants With Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO-MA-MED-0530
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Results first posted 2019-06-28 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2018-06

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Oxymetazoline + Energy-Based Therapy (Experimental): Participants will receive energy-based therapy (Potassium Titanyl Phosphate [KTP], Pulsed Dye Laser [PDL], or Intense Pulsed Light [IPL]) plus once daily application of oxymetazoline hydrochloride (HCl) cream 1.0%.
  Interventions: Drug: Oxymetazoline HCL 1.0% Cream; Device: Energy-Based Therapy

INTERVENTIONS:
Drug: Oxymetazoline HCL 1.0% Cream — Oxymetazoline HCl cream 1.0% once daily application
  Other Names: Rhofade
Device: Energy-Based Therapy — Energy-based therapies (Potassium Titanyl Phosphate [KTP], Pulsed Dye Laser [PDL], or Intense Pulsed Light [IPL])

SUMMARY:
This study will evaluate the safety and tolerability of oxymetazoline HCl cream 1.0% when used as an adjunctive treatment to energy-based therapy for participants with moderate to severe persistent facial erythema associated with rosacea.

ELIGIBILITY:
Inclusion Criteria:

-Documented clinical diagnosis of rosacea.

Exclusion Criteria:

* History of any of the following conditions: Raynaud's syndrome, narrow angle glaucoma, orthostatic hypotension, cerebral or coronary insufficiency, thromboangiitis obliterans, scleroderma, Sjögren's syndrome, severe or unstable or uncontrolled cardiovascular disease, or any other current uncontrolled systemic disease
* Diagnosis or presence of any of the following conditions: rosaceaconglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin, peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or chronic recurring facial acne
* Current treatment with monoamine oxidase (MAO) inhibitors
* Current treatment with niacin ≥ 500 mg/day
* Greater than 3 inflammatory lesions on the face
* History or current evidence of drug or alcohol abuse within 12 months prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Alvandi, Study Director — Allergan
Locations (4):
- United States (4):
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - SkinCare Physicians, Chestnut Hill, Massachusetts
  - Skin Laser and Surgery Specialists of NY/NJ, Hackensack, New Jersey
  - Laser & Skin Surgery Center of New York Professional Corporation, New York, New York

REFERENCES:
- See also: More Information — http://allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxymetazoline + Energy-Based Therapy
Started | 46
Completed | 43
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Oxymetazoline + Energy-Based Therapy
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is defined as any untoward medical occurrence in a clinical study participant administered a medicinal product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not it is related to the medicinal (investigational) product. An SAE is any untoward medical occurrence or effect that, at any dose: Results in death, Is life-threatening, Requires or prolongs inpatient hospitalization, Results in persistent or significant disability/incapacity or Results in a congenital anomaly/birth defect.
Time Frame: Baseline (Day 1) to Day 56
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Oxymetazoline + Energy-Based Therapy
Number analyzed (Participants) | 46
Participants
  TEAES | 5
  Treatment Emergent Serious Adverse Events | 0

2. Primary Outcome: Percentage of Participants With at Least a 1-Grade Improvement From Baseline in the Clinical Erythema Assessment Scale at Any Time-point
Description: The investigator will assess erythema in the treatment area using a 5-point scale. (Grade 0= Clear Skin with no signs of erythema, Grade 1=Almost clear of erythema, slight redness, Grade 2=Mild erythema, definite redness, Grade 3= Moderate erythema, marked redness, Grade 4=Severe erythema, fiery redness). The percentage of participants with at least a 1-point improvement (decrease) in the score compared to Baseline at any time-point will be reported.
Time Frame: Baseline (Day 1) to Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Oxymetazoline + Energy-Based Therapy
Number analyzed (Participants) | 46
Participants
  Day 1 -1 hour post dose | 8
  Day 3-Pre Dose | 21
  Day 3-1 hour post dose | 37
  Day 3-3 hour post dose | 42
  Day 3-6 hour post dose | 37
  Day 3 -post dose any hour | 43
  Day 29 Pre Dose | 18
  Day 29-1 hour post dose | 14
  Day 31 Pre Dose | 26
  Day 31 -1 hour post dose | 38
  Day 31-3 hour post dose | 39
  Day 31-6 hour post dose | 38
  Day 31 -any hour post dose | 42
  Day 56 -Pre Dose | 30
  Day 56-1 hour post dose | 30
  Day 56-3 hour post dose | 40
  Day 56 -6 hour post dose | 39
  Day 56 -any hour post dose | 40

3. Primary Outcome: Percentage of Participants With at Least a 1-Grade Worsening From Baseline in the Clinician's Telangiectasia Assessment (CTA) at Any Time-point
Description: The investigator will assess the overall severity of telangiectasia (spider veins) on the participant's facing using a 5-point scale where 0=Clear skin with no signs of telangiectasia to 4=Severe, with the presence of many visible telangiectasia. The percentage of participants with at least a 1-point worsening (increase) in the score compared to Baseline at any time-point will be reported.
Time Frame: Baseline (Day 1) to Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Oxymetazoline + Energy-Based Therapy
Number analyzed (Participants) | 46
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed the informed consent through Day 56 (Exit Visit)
Arm/Group | Oxymetazoline + Energy-Based Therapy
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 5/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxymetazoline + Energy-Based Therapy (N=46)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 (2)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Pustular (Infections and infestations) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (3)
Face Oedema (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT03380390/SAP_000.pdf
  • Study Protocol (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03380390/Prot_001.pdf